CLINICAL TRIAL: NCT06116708
Title: Effect of the Kalogon AF Prototype Smart Cushion on B52 Pilot Fatigue and Comfort Study
Brief Title: Kalogon Pilot Fatigue and Comfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kalogon (Industry)
Collaborators: EC Service (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 605.019 rev 3
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: B52 Pilot Fatigue and Comfort
Keywords: B52 Pilot; US Air Force; Comfort; Fatigue; Dynamic cushion
MeSH Terms: conditions — Fatigue | interventions — Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 22 Healthy Volunteers (Experimental): Each of the 22 volunteers will participate in a trial with both of the seat cushions. The test order is randomized.
  Interventions: Device: Kalogon AF Prototype Smart Cushion; Device: Standard Seat Cushion from Air Force

INTERVENTIONS:
Device: Kalogon AF Prototype Smart Cushion — The Kalogon cushion is a dynamic smart cushion that utilizes a combination of foam and 5 adjustable air cells to intelligently redistribute weight and increase comfort for users. The air cells are used to modulate interface pressures and adjust where support or pressure reductions are provided based on input from the controller's pressure sensing system.
  Other Names: Kalogon
Device: Standard Seat Cushion from Air Force — This is the standard seat cushion that was provided by the United States Air Force to use for this study. It is a high-density, molded polyurethane foam.
  Other Names: Standard

SUMMARY:
The goal of this experimental study is to compare 2 different seat cushions in B52 cockpit seats to see if they affect pilot fatigue and comfort. The main questions it aims to answer are:

1. Does the Kalogon AF Prototype seat cushion improve pilot comfort compared to the standard seat cushion?
2. Does the Kalogon AF Prototype seat cushion reduce pilot fatigue compared to the standard cushion?

Participants will spend 8 hours in a simulated cockpit playing a flight simulator. They will fill out multiple questionnaires and take 2 attention/reaction time tests throughout the 8-hours.

DETAILED DESCRIPTION:
Participants will be screened for eligibility and if they qualify will be asked to provide informed consent and sign a photo release. Participants will be asked to avoid caffeine consumption on the day of testing, wear comfortable clothing with no back pockets on the pants/shorts, and bring food and water for them to consume during testing.

Once informed consent is given, they will be measured and weighed. They will then be given a flight suit to wear. Once they are in the flight suit, the first 5-minute Psychomotor Vigilance Task test (PVT) will be administered. Once completed, the participant will be strapped into the pilot seat.

Once the participant is properly secured to the pilot seat, the 8-hour timer will be started and the first Subjective Fatigue Survey will be administered. Once the questionnaire is completed they will begin playing the flight simulator. Participants will be encouraged to minimize bathroom breaks and will be given specific times to eat. At the 4-hour mark, the second Subjective Fatigue Survey will be administered. At the end of the 8 hours, a second PVT will be administered, followed by the final Subjective Fatigue Survey.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* 18 to 35 years old
* Ambulatory
* Able to sit for up to 12 hours with minimal breaks
* Able to follow instructions in English

Exclusion Criteria:

* Weight <91 lbs or > 250 lbs
* Pregnant
* Travel across time zones in the last 7 days
* History of:
* Chronic pain
* Asthma or other bronchospasm diagnoses
* Abnormalities of the heart valves, major vessels, heart rate or rhythm, any condition leading to poor circulation, increased risk of blood clots
* Chronic disease of abdominal organs including hepatitis and inflammatory bowel disease
* Un-united fractures, instability of a major joint, retained orthopedic fixation devices, severe scoliosis, or disorder of the skeletal muscles
* Psoriasis
* Psychosis, schizophrenia, or other severe mental health disorder
* Seizure disorders
* Sleeping disorders
* Taking any of the following medications:
* Opiates
* Muscle relaxants
* Anticholinergics
* Sedating antihistamines
* Anti-psychotics

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Comfort | Beginning of trial (T0), 4 hours into the trial (T1), and at the end of the trial (T2), 8 hours after T0.
  The subjective measure of the amount of discomfort and comfort that a participant experiences from sitting on the cushions. This outcome is evaluated using a Subjective Fatigue Survey that has 2 parts. The first part is a 35 question Discomfort Assessment that utilizes a labeled body map to allow volunteers to rate their level of discomfort in each body zone. The second part of the Subjective Fatigue Survey is a 13 question Comfort Assessment that contains 13 statements on the topic of comfort that volunteers indicate how much they agree with that statement using an 11-point Likert scale.
Fatigue | Beginning of the trial (T0) and at the end (T2), 8 hours apart.
  A psychomotor vigilance task test is utilized to measure fatigue through changes in response time.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Call, MS, CSM-NRM, Principal Investigator — EC Service
Locations (1):
- Kalogon Headquarters, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, the protocol and report will be made available to the Air Force Research Lab (AFRL) for their review.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The CSR will be made available no later than December 15, 2023. The ICF, SAP, and study protocol were provided to them prior to the initiation of the study.
Access Criteria: All data will be deidentified and will be available to designated personnel at the AFRL

REFERENCES:
- [Background] Arsintescu L, Kato KH, Cravalho PF, Feick NH, Stone LS, Flynn-Evans EE. Validation of a touchscreen psychomotor vigilance task. Accid Anal Prev. 2019 May;126:173-176. doi: 10.1016/j.aap.2017.11.041. Epub 2017 Dec 2. PMID 29198969
- [Background] Vanacore A, Lanzotti A, Percuoco C, Capasso A, Vitolo B. Design and analysis of comparative experiments to assess the (dis-)comfort of aircraft seating. Appl Ergon. 2019 Apr;76:155-163. doi: 10.1016/j.apergo.2018.12.012. Epub 2019 Jan 8. PMID 30642520
- [Background] Shen W, Parsons KC. Validity and reliability of rating scales for seated pressure discomfort. International Journal of Industrial Ergonomics. 1997; 20(6), 441-461
- See also: FAA Medications List — https://www.faa.gov/ame_guide/media/DNI_DNF_tables.pdf
- See also: Air Force Weight Requirements — https://www.military.com/military-fitness/air-force-fitness-requirements/air-force-height-and-weight-charts

DOCUMENTS (2):
  • Study Protocol (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT06116708/Prot_001.pdf
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT06116708/ICF_002.pdf